CLINICAL TRIAL: NCT03499912
Title: Screening of IDH1 and IDH2 Gene Mutations in Adult Acute Myeloid Leukemia for Possible Targeted Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201701030RIPC
Record Dates: First submitted 2018-03-22; First posted 2018-04-17 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; IDH1; IDH2; Genetic mutations; Prognosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. To assess the incidence of IDH1 and IDH2 mutations in adult AML patients, and to explore their associations with the patients' clinical, cytogenetic, and molecular characteristics as well as with treatment response and outcome.
2. To delineate the similarities and distinctions among mutations at IDH1-R132, IDH2-R140 and IDH2-R172 in AML, both clinically and molecularly (including cytogenetics, immunophenotyping, mutation co-occurrence patterns).
3. The results can be references for future selection of targeted therapy (targeting IDH mutant proteins).

DETAILED DESCRIPTION:
Isocitrate dehydrogenases (IDH) are enzymes that catalyze oxidative decarboxylation of isocitrate into alpha-ketoglutarate (α-KG). IDH1 and IDH2 mutations in AML give the enzymes neomorphic enzymatic activity to transform α-KG to D-2HG, an oncometabolite which acts as a competitive inhibitor of dioxygenases, and causes dysregulation of TET2 and histone demethylases, consequently leading to epigenetic reprogramming of a cell, blocking differentiation and contributing to a transformed phenotype, and leukemogenesis. Investigators plan to recruit 300 adult AML patients (newly diagnosed or relapsed). 10mL of peripheral blood or marrow blood will be obtained from routine practice blood/marrow sampling specimens (no extra venipuncture or bone marrow aspiration would be required) and sent for routine tests such as cytogenetics, immunophenotyping, and gene mutation analyses. IDH1 R132, IDH2 R140, and IDH2 R172 mutations will be screened by PCR followed by Sanger sequencing, as previously described.

Investigators will first assess the incidence of IDH1 and IDH2 mutations in adult AML patients, and then explore their associations with the patients' clinical course, cytogenetic, and molecular characteristics as well as with treatment response and outcome. Investigators also seek to delineate the similarities and distinctions among IDH mutation variants at IDH1-R132, IDH2-R140 and IDH2-R172, both clinically and molecularly (including cytogenetics, immunophenotyping, mutation co-occurrence patterns).

ELIGIBILITY:
Inclusion criteria:

1. Patients ≥20 Years with Diagnosed Acute Myeloid Leukemia
2. Willing to provide voluntary written informed consent before study related procedures

Exclusion criteria:

1. Not acute myeloid leukemia patients
2. Patients <20 Years with Diagnosed Acute Myeloid Leukemia

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult AML patients (newly diagnosed or relapsed) diagnosed at the National Taiwan University Hospital (NTUH) according to the updated 2016 WHO AML classification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of IDH1 and IDH2 mutation | 2017/03/07 - 2019/03/01
  Peripheral blood or marrow blood will be obtained from routine practice blood/marrow sampling specimens (no extra venipuncture or bone marrow aspiration would be required) and sent for routine tests such as cytogenetics, immunophenotyping, and gene mutation analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chien Chou, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan